CLINICAL TRIAL: NCT02357199
Title: Interventional Study Targeting Oral Infections in Patients With Chronic Kidney Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: Rigshospitalet, Denmark (Other); Danish Council for Independent Research - Medical Sciences (Unknown); The Danish Dental Association (Unknown)
Responsible Party: Principal Investigator, Siri Beier Jensen, Associate Professor, DDS, PhD, University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 102-2084/14-3000
Record Dates: First submitted 2015-01-28; First posted 2015-02-06 (Estimated); Last update posted 2015-08-31 (Estimated); Status verified 2015-08

CONDITIONS: Mouth Diseases; Renal Insufficiency, Chronic
Keywords: Mouth Diseases; Renal Insufficiency, Chronic; Intervention Studies
MeSH Terms: conditions — Mouth Diseases; Renal Insufficiency, Chronic

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intensive oral care & didactic training (Experimental): Professional (dental hygienist) intensive oral care intervention and individual patient training/didactic instruction to promote patient compliance and patient capability of oral preventive measures in a long-term perspective.
  Interventions: Other: Intensive oral care & didactic training
- Standard oral care (No Intervention): Standard oral care protocol consisting of referral by staff in the Department of Nephrology to general dental practitioner followed by patient self-administration of tooth brushing, fluoride toothpaste and oral lubricants.

INTERVENTIONS:
Other: Intensive oral care & didactic training — Professional (dental hygienist) intensive oral care intervention and individual patient training/didactic instruction to promote patient compliance and patient capability of oral preventive measures in a long-term perspective.
  Arms: Intensive oral care & didactic training

SUMMARY:
This study aims to investigate the prevalence of oral infection in chronic renal disease patients and to examine whether a focused oral hygiene intervention can reduce oral infection leading to reduced systemic inflammatory parameters in chronic renal disease patients in hemodialysis, chronic renal disease patients waiting for kidney transplantation, and chronic renal disease patients who has been transplanted 1-1½ year previously. The results will be compared to a gender- and age-matched healthy control group.

DETAILED DESCRIPTION:
Aim:

The aim is to examine if a focused oral care procedure to reduce oral infection will be mirrored in reduction of systemic inflammatory parameters in chronic renal disease patients.

Specific research questions:

Can oral infection and systemic inflammatory parameters in chronic renal disease patients be reduced by 1 month of professional oral care and individual prophylactic instruction and can a potential reduction of inflammation be continuously achieved at a 3 months follow-up.

Study design:

Randomized, double-blinded (investigator, outcomes assessor), controlled study. For Eligibility Criteria and Outcome Measures, please see elsewhere in the ClinicalTrials.gov Protocol Registration System.

Participants:

A: Hemodialysis patients, inclusion n=34, B: Hemodialysis patients on a kidney transplant waiting list, inclusion n=34, C: Patients who have had a kidney transplant (1-1½ years after transplantation), inclusion n=34. D: Gender- and age-matched healthy control group.

Number of included patients is estimated from a hypothesis-generating pilot study, a statistical power analysis and the estimated loss to follow-up based on experience from previous research projects in the Nephrology Department.

Intervention and control:

The intervention consists of professional oral care (addressing periodontal and oral mucosal infections, salivary gland dysfunction and caries prevention) and a didactic approach to individual instruction in oral hygiene/prophylactic measures performed by a dental hygienist at three visits: baseline, 2 weeks after baseline and 1 month after baseline.

The research data will be registered by a blinded investigator before the first visit at the dental hygienist and after 3 months.

The control group will follow best-clinical-practice procedures currently implemented in the hospital.

ELIGIBILITY:
Inclusion Criteria:

* Patients on a kidney transplant waiting list or patients who have had a kidney transplant (1-1½ year previously)
* Dentate patients (>10 teeth)
* Age >18 years
* Danish language

Exclusion Criteria:

* Patients not capable of following the research protocol
* Legally unavailable
* Need of antibiotic prophylaxis with dental treatment
* Heart valve surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2015-01; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Gingival inflammation | Change from baseline examination (before oral care intervention) at 3-months follow-up examination
  Gingival inflammation measured by gingivitis index
C-reactive protein, plasma | Change from baseline examination (before oral care intervention) at 3-months follow-up examination
  Blood sample

SECONDARY OUTCOMES:
Dental bacterial plaque | Change from baseline examination (before oral care intervention) at 3-months follow-up examination
  Measured by plaque index
Periodontal disease | Change from baseline examination (before oral care intervention) at 3-months follow-up examination
  Measurement of attachment level
Whole saliva flow rate, unstimulated | Change from baseline examination (before oral care intervention) at 3-months follow-up examination
  Sialometry
Whole saliva flow rate, stimulated | Change from baseline examination (before oral care intervention) at 3-months follow-up examination
  Sialometry
Saliva composition: Sodium | Change from baseline examination (before oral care intervention) at 3-months follow-up examination
  Sialochemistry
Saliva composition: Chloride | Change from baseline examination (before oral care intervention) at 3-months follow-up examination
  Sialochemistry
Saliva composition: Potassium | Change from baseline examination (before oral care intervention) at 3-months follow-up examination
  Sialochemistry
Saliva composition: Total calcium | Change from baseline examination (before oral care intervention) at 3-months follow-up examination
  Sialochemistry
Saliva composition: Inorganic phosphate | Change from baseline examination (before oral care intervention) at 3-months follow-up examination
  Sialochemistry
Saliva composition: Total protein | Change from baseline examination (before oral care intervention) at 3-months follow-up examination
  Sialochemistry
Saliva composition: Albumin | Change from baseline examination (before oral care intervention) at 3-months follow-up examination
  Sialochemistry
Saliva composition: Amylase activity | Change from baseline examination (before oral care intervention) at 3-months follow-up examination
  Sialochemistry
Saliva composition: Secretory IgA | Change from baseline examination (before oral care intervention) at 3-months follow-up examination
  Sialochemistry
Oral candidiasis | Change from baseline examination (before oral care intervention) at 3-months follow-up examination
  Smear test
Hematologic status: Erythrocytes | Change from baseline examination (before oral care intervention) at 3-months follow-up examination
  Blood sample
Hematologic status: Hemoglobin | Change from baseline examination (before oral care intervention) at 3-months follow-up examination
  Blood sample
Hematologic status: Leukocytes | Change from baseline examination (before oral care intervention) at 3-months follow-up examination
  Blood sample
Hematologic status: Thrombocytes | Change from baseline examination (before oral care intervention) at 3-months follow-up examination
  Blood sample
Hematologic status: Transferrin | Change from baseline examination (before oral care intervention) at 3-months follow-up examination
  Blood sample
Hematologic status: Iron | Change from baseline examination (before oral care intervention) at 3-months follow-up examination
  Blood sample
Calcium metabolism | Change from baseline examination (before oral care intervention) at 3-months follow-up examination
  Blood sample
Phosphate metabolism | Change from baseline examination (before oral care intervention) at 3-months follow-up examination
  Blood sample
Renal function: Carbamide | Change from baseline examination (before oral care intervention) at 3-months follow-up examination
  Blood sample
Renal function: Bicarbonate | Change from baseline examination (before oral care intervention) at 3-months follow-up examination
  Blood sample
Renal function: Creatinine | Change from baseline examination (before oral care intervention) at 3-months follow-up examination
  Blood sample
Renal function: Albumin | Change from baseline examination (before oral care intervention) at 3-months follow-up examination
  Blood sample
Renal function: Potassium | Change from baseline examination (before oral care intervention) at 3-months follow-up examination
  Blood sample
Renal function: Sodium | Change from baseline examination (before oral care intervention) at 3-months follow-up examination
  Blood sample
Oral Health Impact Profile | Change from baseline examination (before oral care intervention) at 3-months follow-up examination
  Quality of life questionnaire
Medical Outcomes Study Short Version | Change from baseline examination (before oral care intervention) at 3-months follow-up examination
  Quality of life questionnaire

OTHER OUTCOMES:
Dental caries | Baseline examination (before oral care intervention), 3-months follow-up examination
  Clinical registration of dental caries

CONTACTS AND LOCATIONS:
Overall Officials: Siri B Jensen, DDS, PhD, Principal Investigator — University of Copenhagen
Locations (1):
- Department of Odontology, Faculty of Health Sciences, University of Copenhagen, Copenhagen, Denmark

REFERENCES:
- [Background] Kato S, Chmielewski M, Honda H, Pecoits-Filho R, Matsuo S, Yuzawa Y, Tranaeus A, Stenvinkel P, Lindholm B. Aspects of immune dysfunction in end-stage renal disease. Clin J Am Soc Nephrol. 2008 Sep;3(5):1526-33. doi: 10.2215/CJN.00950208. Epub 2008 Aug 13. PMID 18701615
- [Background] McIntyre C, Harper I, Macdougall IC, Raine AE, Williams A, Baker LR. Serum C-reactive protein as a marker for infection and inflammation in regular dialysis patients. Clin Nephrol. 1997 Dec;48(6):371-4. PMID 9438096
- [Background] Thorman R. Oral health in patients with chronic kidney disease. Stockholm, Sweden: Karolinska Institutet; 2009